CLINICAL TRIAL: NCT02816112
Title: A Multi-Centre Study to Compare Granulocyte-colony Stimulating Factors to Antibiotics for Primary Prophylaxis of Taxotere/Cyclophosphamide-Induced Febrile Neutropenia REaCT-TC2
Brief Title: Granulocyte-colony Stimulating Factors or Antibiotics for Primary Prophylaxis for Febrile Neutropenia
Acronym: REaCT-TC2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTT 16-03
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Early Stage Breast Cancer
MeSH Terms: interventions — Ciprofloxacin; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ciprofloxacin (Active Comparator): Oral tablet taken twice a day at home starting 5 days after chemotherapy for 14 days for every cycle of TC
  Interventions: Drug: Ciprofloxacin
- G-CSF (Active Comparator): Daily injection at home for the number of days as chosen by the treating physician
  Interventions: Drug: Neupogen

INTERVENTIONS:
Drug: Ciprofloxacin — Antibiotic
  Arms: Ciprofloxacin
Drug: Neupogen — Granulocyte-colony stimulating factor
  Other Names: filgrastim
  Arms: G-CSF

SUMMARY:
Taxotere-cyclophosphamide (TC) chemotherapy is commonly used as an adjuvant chemotherapy regimen in patients with resected early stage breast cancer. TC chemotherapy can cause febrile neutropenia (FN) which can be serious and associated with treatment delays and dose reductions, thereby compromising treatment efficacy. To reduce the risk of chemotherapy-induced FN,TC is administered with either one of two highly effective standard treatments; namely primary prophylaxis with either ciprofloxacin or granulocyte colony-stimulating factor (G-CSF). However, there are considerable cost differences between these strategies; subcutaneous daily G-CSF costs at least $12,000 over 4 cycles of treatment while oral ciprofloxacin costs about $100.

The investigators have therefore been performing a feasibility study to explore whether the "integrated consent model" involving oral consent is feasible in practice; and whether it can be used to increase the number of physicians and patients who take part in clinical trials. This feasibility study (REaCT-TC NCT02173262) has been an amazing success and the investigators are therefore now performing a definitive study comparing G-CSF with ciprofloxacin. This study will not be evaluating feasibility endpoints, but rather clinically important endpoints of hospitalizations and febrile neutropenia rates.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary breast cancer
* Planned TC chemotherapy
* ≥19 years of age
* Able to provide verbal consent

Exclusion Criteria:

* Contraindication to either Ciprofloxacin or G-CSF

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2016-09; Primary Completion 2020-03 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Febrile neutropenia | 2 years
  Number of participants with febrile neutropenia
Treatment-related hospitalization | 2 years
  Number of participants admitted to hospital for treatment-related reasons

SECONDARY OUTCOMES:
Chemotherapy dose reduction | 2 years
  Number of participants who receive a dose reduction of their TC chemotherapy
Chemotherapy dose delay | 2 years
  Number of participants who receive a dose delay in their TC chemotherapy
Chemotherapy discontinuation | 2 years
  Number of participants who stop TC chemotherapy for any reason
Microbiologic infections | 2 years
  Number of participants who have a microbiologic infection (i.e: Clostridium difficile)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clemons, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IDP available.